CLINICAL TRIAL: NCT04951778
Title: A Phase 1, Open-label, Dose-finding Study of CC-91633 (BMS-986397) in Subjects With Relapsed or Refractory Acute Myeloid Leukemia or Relapsed or Refractory Higher-Risk Myelodysplastic Syndromes
Brief Title: Study to Evaluate Safety and Tolerability of CC-91633 (BMS-986397) in Participants With Relapsed or Refractory Acute Myeloid Leukemia or Relapsed or Refractory Higher-Risk Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Efficacy endpoint met; however, overall experimental dosing regimen is not considered optimal to support further clinical development in this patient population
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CC-91633-AML-001; 2020-005329-95 (EudraCT Number)
Record Dates: First submitted 2021-06-23; First posted 2021-07-07 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
Keywords: Relapsed or Refractory Acute Myeloid Leukemia; Relapsed or Refractory Higher-Risk Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Participants with R/R AML and R/R HR-MDS - Part A (Experimental): Part A (Dose Escalation) of the study will enroll R/R AML (Relapsed or Refractory Acute Myeloid Leukemia) and R/R HR-MDS (Relapsed or Refractory Higher-Risk Myelodysplastic Syndromes) participants and will evaluate the safety and tolerability of escalating doses of CC-91633, administered orally, and determine the maximum tolerated dose (MTD) or preliminary recommended Phase 2 doses (RP2D) and schedule.
  Interventions: Drug: CC-91633
- Participants with Relapsed or Refractory Acute Myeloid Leukemia (R/R AML) (Experimental): Part B (expansion part) will confirm tolerability of the selected doses and schedules and evaluate whether efficacy is in a range that warrants further clinical development for R/R AML participants.
  Interventions: Drug: CC-91633
- Participants with Relapsed or Refractory Higher-Risk Myelodysplastic Syndromes (HR-MDS) (Experimental): Part B (expansion part) will confirm tolerability of the selected doses and schedules and evaluate whether efficacy is in a range that warrants further clinical development for R/R HR-MDS participants.
  Interventions: Drug: CC-91633

INTERVENTIONS:
Drug: CC-91633 — Administered orally according to the assigned treatment schedule
  Other Names: BMS-986397

SUMMARY:
Study CC-91633-AML-001 is a Phase 1, open-label, dose escalation and expansion, first-in-human (FIH) clinical study of CC-91633 (BMS-986397) in participants with relapsed or refractory acute myeloid leukemia (R/R AML) or in participants with relapsed or refractory higher-risk myelodysplastic syndromes (R/R HR-MDS). The Dose Escalation part (Part A) of the study will enroll participants with R/R AML and R/R HR-MDS and will evaluate the safety and tolerability of escalating doses of CC-91633 (BMS-986397), administered orally, and determine the maximum tolerated dose (MTD) or preliminary recommended Phase 2 doses (RP2D) and schedule. Throughout the study, final decisions on dose escalation/de-escalation will be made by the safety review committee (SRC). Approximately 60 participants may be enrolled in Part A of the study.

The expansion part (Part B) will confirm tolerability of the selected doses and schedules and evaluate whether efficacy is in a range that warrants further clinical development. Approximately 60 response-evaluable subjects per indication (R/R AML or R/R HR-MDS) may be enrolled.

Parts A and B will consist of 3 periods: Screening, Treatment, and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the criteria below to be enrolled in the Dose Escalation (Part A) or the Dose Expansion (Part B) of this study.

* Participant is ≥ 18 years of age, at the time of signing the ICF.
* Participant must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
* Participant is willing and able to adhere to the study visit schedule and other protocol requirements.
* Relapsed or refractory acute myeloid leukemia (R/R AML) and relapsed or refractory higher-risk myelodysplastic syndromes (R/R HR-MDS) as defined by the World Health Organization (WHO) criteria who have failed or are ineligible for all available therapies which may provide clinical benefit
* Participant has Eastern Cooperative Oncology Group Performance Status of 0 to 2.
* Participants must have the following screening laboratory values:

  * Total White Blood Cell count (WBC) < 25 x 109/L prior to first infusion.
  * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 3.0 x upper limit of normal (ULN), unless considered due to leukemic organ involvement, in which case AST and ALT can be ≤ 5.0 x ULN.
  * Uric acid ≤ 7.5 mg/dL (446 μmol/L).
  * Serum total bilirubin ≤ 1.5 x ULN, unless considered due to Gilbert's syndrome
  * Estimated serum creatinine clearance of ≥ 60 mL/min using the Cockcroft-Gault equation. Measured creatinine clearance from a 24-hour urine collection is acceptable if clinically indicated.
  * INR < 1.5 x ULN and partial thromboplastin time (PTT) < 1.5 x ULN.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

* Participant has any condition, including active or uncontrolled infection, or the presence of laboratory abnormalities, which places the participant at unacceptable risk if the participant were to participate in the study.
* Any other significant medical condition, laboratory abnormality, or psychiatric illness which places the participant at unacceptable risk if he/she were to participate in the study or that would prevent the participant from complying with the study.
* Participant has any condition that confounds the ability to interpret data from the study.
* Participants with acute promyelocytic leukemia.
* Participants with clinical symptoms suggesting active central nervous system (CNS) leukemia or known CNS leukemia.
* Participants with immediately life-threatening, severe complications of leukemia such as disseminated/uncontrolled infection, uncontrolled bleeding, and/or uncontrolled disseminated intravascular coagulation.
* Participants with impaired cardiac function or clinically significant cardiac diseases,
* Participants who have undergone major surgery ≤ 2 weeks prior to starting CC-91633. Participants must have recovered from any clinically significant effects of recent surgery.
* Pregnant or nursing individuals.
* Participants with known human immunodeficiency virus infection.
* Participants with known chronic, active hepatitis B virus or hepatitis C virus C (HCV) infection.
* Participants with ongoing treatment with chronic, therapeutic dosing of anticoagulants (eg, warfarin, low molecular weight heparin, Factor Xa inhibitors).
* Participants with history of concurrent second cancers requiring active, ongoing systemic treatment
* Participants with clinically significant diarrhea, vomiting or malabsorption felt to limit absorption of orally administered medications.
* Participants with known or suspected hypersensitivity to any of the components or excipients of the study treatment or to similar class drugs (eg, lenalidomide).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 2 years
  Defined as the dose with highest posterior probability of the Dose-limiting toxicity (DLT) rate falling in the target interval and fulfilling escalation with overdose control (EWOC).
Dose-limiting Toxicity (DLT) | Up to 42 days after first dose of study treatment in Part A
  Defined as toxicities such as non-hematologic, confirmed Hy's law case, hematologic, or any AE toxicities meeting protocol specified DLT criteria and occurring within the DLT assessment period, unless the toxicity can clearly be determined to be due to other specified causes.
Incidence of Adverse Events (AEs) | Up to 4 years
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

SECONDARY OUTCOMES:
Complete Remission Rate (CRR) | Up to 4 years
  Complete remission rate (CRR) is defined as the percent of participants whose best response is CRs including complete remission (CR), complete remission with partial hematologic recovery (CRh) and complete remission with incomplete hematologic recovery (CRi).
Efficacy determined by response rates of Acute Myeloid Leukemia (AML) - Minimal residual disease negative complete remission rate (CRRMRD-) | Up to 4 years
  Minimal residual disease negative complete remission rate is defined as the percent of participants with Minimal residual disease negative complete remission.
Efficacy determined by response rates of Acute Myeloid Leukemia (AML) - Combined Complete Remission Rate (cCRR) | Up to 4 years
  Combined complete remission rate (cCRR), is defined as the percent of participants whose best response is complete remission, includes minimal residual disease negative complete remission rate (CRRMRD-), morphologic complete remission, complete remission with incomplete hematologic recovery (CRi), complete remission with partial hematologic recovery (CRh).
Efficacy determined by response rates of Acute Myeloid Leukemia (AML) - Morphologic Leukemia-free State Rate (MLFSR) | Up to 4 years
  The Morphologic Leukemia-free State Rate is defined as the percent of participants with the best response of Morphologic Leukemia-free State.
Partial Remission Rate (PRR) | Up to 4 years
  Partial Remission Rate is defined as the percent of participant with the best response of Partial Remission.
Stable Disease Rate (SDR) | Up to 4 years
  Stable Disease Rate is defined as the percent of participants with the best response of Stable Disease.
Progression-free Survival (PFS) rate at 3 and 9 months | At 3 months and 9 months of PFS
  Progression free survival rate is defined as the percent of participants with progression free for at least 3/9 months.
Overall Survival (OS) rate | At 6 and 12 months of survival
  Overall survival rate is defined as the percent of participant who have survived for at least 6/12 months.
Overall Response Rate (ORR) | Up to 4 years
  Overall response rate is defined as the percent of participants whose best response is any of those composite complete response rate (cCRR) or morphologic Leukemia-free state (MLFS) or partial remission (PR) for AML and any of CR, marrow CR with HI (mCRHIR), PR, hematologic improvement (HI) for MDS.
Overall Survival (OS) | Up to 4 years
  Overall Survival is measured as the time from the first dose of CC-91633 to death due to any cause.
Relapse-free Survival (RFS) | Up to 4 years
  Relapse-free survival is defined only for participants who have achieved the best response of any of CR/CRh/CRi/CRRMRD- or any of PR/MLFS/mCRHIR/HI, and is measured as the interval from the date of first achieved of any CR/CRh/Cri/CRRMRD- or any of PR/ MLFS/mCRHIR/HI to the date of disease relapse or death from any cause, whichever occurs first.
Progression-free Survival (PFS) | Up to 4 years
  Progression-Free Survival is defined as the time from the first dose of CC-91633 to the first occurrence of relapse or progression or death from any cause.
Event-free Survival (EFS) | Up to 4 years
  Event-free Survival is defined as the interval from the date of the first dose to an event including disease progression, treatment failure, relapse, or death from any cause, whichever occurs first.
Duration of remission/response | Up to 4 years
  For participants with best response of any of CR/CRh/ CRi/CRRMRD- or any of PR/MLFS/mCRHIR/HI, duration of remission/response is measured from the time when criteria for the best response of any of CR/CRh/ Cri/CRRMRD- or any of PR/ MLFS/mCRHIR/HI are first met (whichever is first recorded) until the first date at which relapse, or progressive disease is objectively documented assessment.
Time to remission/response | Up to 4 years
  Time to onset of first remission/response is defined as the time interval from the date of first dose and the earliest date any remission/response (any CRs or PR) is observed.
Efficacy: Time to transformation to Acute Myeloid Leukemia (AML) for High-Risk Myelodysplastic Syndrome (HR-MDS) | Up to 4 years
  Time interval from first dose to onset date of having 20% more bone marrow (BM) or peripheral blood (PB) blasts.
CC-91633 Pharmacokinetics - Cmax | Up to 4 years
  Maximum plasma drug concentration.
CC-91633 Pharmacokinetics - AUC(0-T) | Up to 4 years
  Area under the plasma concentration-time curve from time zero to time t, where t is the time point of the last measurable concentration.
CC-91633 Pharmacokinetics - AUC(TAU) | Up to 4 years
  Area under the plasma concentration time-curve from time 0 to 24 hours postdose.
CC-91633 Pharmacokinetics - Tmax | Up to 4 years
  Time to peak (maximum) plasma concentration.
CC-91633 Pharmacokinetics - T-HALF | Up to 4 years
  Half-life.
CC-91633 Pharmacokinetics - CLT/F | Up to 4 years
  Apparent total clearance of the drug from plasma after oral administration, as appropriate.
CC-91633 Pharmacokinetics - Vz/F | Up to 4 years
  Apparent volume of distribution, as appropriate.
CC-2004772 Pharmacokinetics - Cmax | Up to 4 years
  Maximum plasma drug concentration, if possible.
CC-2004772 Pharmacokinetics - AUC(0-T) | Up to 4 years
  Area under the plasma concentration-time curve from time zero to time t, where t is the time point of the last measurable concentration, if possible.
CC-2004772 Pharmacokinetics - AUC(TAU) | Up to 4 years
  Area under the plasma concentration time-curve from time 0 to 24 hours postdose, if possible.
CC-2004772 Pharmacokinetics - Tmax | Up to 4 years
  Time to peak (maximum) plasma concentration, if possible.
CC-2004772 Pharmacokinetics - T-HALF | Up to 4 years
  Half-life, if possible.
CC-2004772 Pharmacokinetics - CLT/F | Up to 4 years
  Apparent total clearance of the drug from plasma after oral administration, if possible.
CC-2004772 Pharmacokinetics - Vz/F | Up to 4 years
  Apparent volume of distribution, if possible.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (5):
  - Local Institution - 107, Boston, Massachusetts
  - Local Institution - 101, Boston, Massachusetts
  - Local Institution - 105, St Louis, Missouri
  - Local Institution - 104, Houston, Texas
  - Local Institution - 109, Seattle, Washington
- Spain (4):
  - Local Institution - 302, Barcelona
  - Local Institution - 301, Barcelona
  - Local Institution - 303, Madrid
  - Local Institution - 304, Seville

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com